CLINICAL TRIAL: NCT01276990
Title: Safety and Pharmacokinetics of Multiple Rising Oral Doses of BI 224436 ZW (Powder in Bottle Formulation) at 12.5 mg q24h, 12.5 mg q12h, 12.5 mg q8h, 25 mg q12h, 25 mg q8h, 50 mg q12h, 37.5 mg q8h and 50 mg q8h Dose Levels for 10 Days in Healthy Male Volunteers (Randomized, Double-blind Placebo-controlled Within Dose Groups)
Brief Title: Safety and Pharmacokinetics of Multiple Rising Oral Doses of BI 224436 in Healthy Male Volunteers.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1277.2
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: HIV Infections; Healthy
MeSH Terms: conditions — HIV Infections

ARMS (9):
- Placebo (Placebo Comparator): Matching placebo in dosing regimen 1-8
  Interventions: Drug: BI 224436; Drug: Placebo
- BI 224436 dosing regimen 1 (Experimental): Dosing regimen 1
  Interventions: Drug: BI 224436
- BI 224436 dosing regimen 2 (Experimental): Dosing regimen 2
  Interventions: Drug: BI 224436
- BI 224436 dosing regimen 3 (Experimental): Dosing regimen 3
  Interventions: Drug: BI 224436
- BI 224436 dosing regimen 4 (Experimental): Dosing regimen 4
  Interventions: Drug: BI 224436
- BI 224436 dosing regimen 5 (Experimental): Dosing regimen 5
  Interventions: Drug: BI 224436
- BI 224436 dosing regimen 6 (Experimental): Dosing regimen 6
  Interventions: Drug: BI 224436
- BI 224436 dosing regimen 7 (Experimental): Dosing regimen 7
  Interventions: Drug: BI 224436
- BI 224436 dosing regimen 8 (Experimental): Dosing regimen 8
  Interventions: Drug: BI 224436

INTERVENTIONS:
Drug: BI 224436 — Oral drinking solution
  Arms: BI 224436 dosing regimen 6
Drug: BI 224436 — Oral drinking solution
  Arms: BI 224436 dosing regimen 8
Drug: BI 224436 — Oral drinking solution
  Arms: BI 224436 dosing regimen 2
Drug: BI 224436 — Oral drinking solution
  Arms: BI 224436 dosing regimen 3
Drug: BI 224436 — Oral drinking solution
  Arms: BI 224436 dosing regimen 4
Drug: BI 224436 — Oral drinking solution
  Arms: BI 224436 dosing regimen 5
Drug: BI 224436 — Oral drinking solution
  Arms: BI 224436 dosing regimen 7
Drug: BI 224436 — Oral drinking solution
  Arms: Placebo
Drug: BI 224436 — Oral drinking solution
  Arms: BI 224436 dosing regimen 1
Drug: Placebo — Oral drinking solution
  Arms: Placebo

SUMMARY:
To investigate the safety and pharmacokinetic of BI 224436 in healthy male volunteers following oral administration of repeated doses for 10 days within 8 dosing regimens.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male according to the following criteria: based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests.
2. Age >=18 and <=50 years.
3. Body Mass Index (BMI) >=18.5 and BMI <=32 kg/m2.
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation.
5. Documented to be sterile; or, if can father a child, agree to abstain from sexual intercourse during and at least seven days following last study drug administration, or are willing to use condoms during the same period each time (Subject's female sexual partner(s) of child-bearing potential should be willing to use either ethinyl estradiol containing oral contraceptives or a reliable barrier method of contraception).

Exclusion criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance according to the opinion of the investigator.
2. Any evidence of a clinically relevant concomitant disease.
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
4. Surgery of the gastrointestinal tract that in the opinion of the investigator may affect the absorption.
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders.
6. History of relevant orthostatic hypotension, fainting spells or blackouts.
7. History or evidence of Human Immunodeficiency Virus or other chronic or relevant acute infections, including Hepatitis C Virus and Hepatitis B Virus infection.
8. History of relevant allergy / hypersensitivity (including allergy to investigational medicinal product or its solvent).
9. History of any familial skeletal muscle disorder, or history of Creatine Kinase (CK) elevation not due to strenuous physical activity or trauma.
10. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial.
11. Use of drugs, including prescription and non-prescription drugs, and St. Johns Wort which might reasonably influence the results of the trial within 14 days prior to study drug administration or during the trial, or consumption of grapefruit, grapefruit juice, orange juice, Seville oranges, green tea, pineapple, pineapple juice, broccoli or red wine within 3 days prior study drug administration or during the trial.
12. Participation in another trial with an investigational drug within one month prior to administration or during the trial.
13. Current smoker (>10 cigarettes or >3 cigars or >3 pipes / day).
14. Inability to refrain from smoking during the trial.
15. Alcohol abuse (more than 30 g day).
16. Drug abuse.
17. Blood donation (more than 100 mL within four weeks prior to administration or during the trial).
18. Physical activity in excess of usual activity of daily living (e.g., fitness physical exercise, physical labor) within 7 days prior to study drug administration until end of study visit.
19. Any laboratory value outside the reference range that in the opinion of the investigator is of clinical relevance.
20. A marked baseline prolongation of QT or corrected QT (QTc) intervals (e.g., repeated demonstration of a QTc interval >450 ms); or, other ECG abnormality of clinical significance.
21. A history of additional risk factors for Torsades de points (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
22. CK at screening =2x Upper Limit of Normal (ULN) (If CK is =2xULN and <5xULN one retest will be allowed to verify the result).
23. CK at baseline (Day -1) >ULN (If CK is >ULN and <1.5xULN one retest will be allowed to verify the result).
24. Thyroid - stimulating hormone outside normal reference range, or history of hypo-or hyperthyroidism.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Changes in blood pressure | 1 month
Changes in pulse rate | 1 month
Changes in 12-lead ECG | 1 month
Changes in clinical laboratory test parameters | 1 month
Adverse events | 1 month

SECONDARY OUTCOMES:
Cmax,ss (maximum measured concentration of the analyte in plasma at steady-state over a uniform dosing interval t) | 10 days
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady-state) | 10 Days
Cmin,ss (minimum concentration of the analyte in plasma at steady-state over a uniform dosing interval t) | 10 days
AUCt,ss (area under the concentration-time curve of the analyte in plasma at steady-state over a uniform dosing interval t) | 13 days
t1/2,ss (terminal half-life of the analyte in plasma at steady-state) | 13 days
CL/F,ss (apparent clearance of the analyte in the plasma at steady-state following extravascular multiple dose administration) | 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim